CLINICAL TRIAL: NCT02539953
Title: Ambulatory Blood Pressure Monitoring in Rivaroxaban Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KCH1002
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2015-02

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring — Patients with dizziness on taking rivaroxaban will have ambulatory blood pressure monitoring to assess haemodynamic effects indirectly

SUMMARY:
One in ten patients on rivaroxaban therapy have dizziness and reductions in blood pressure. The investigators intend to monitor the ambulatory blood pressure of such patients in order to assess whether this is a true haemodynamic effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Able to provide written, informed consent
* Taking rivaroxaban for any indication within the license of the drug, both once daily and twice daily dosing can be included
* Have measurable rivaroxaban levels on at least one occasion (this will be in line with standard of care, there will be no extra blood samples for the study)
* Not taking concomitant medication that can affect rivaroxaban metabolism (including amiodarone, dronedarone, -azole antifungals, protease inhibitors)
* On no antihypertensive or vasoactive medication
* Have a baseline BP recording taken in clinic

Exclusion Criteria:

* Unable to provide written, informed consent
* Presence of concomitant medication that may alter rivaroxaban levels and confound results (see above)
* Unwilling to undergo ambulatory blood pressure monitoring
* Contraindication to ambulatory blood pressure monitoring

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Average blood pressure readings | 48 hours

SECONDARY OUTCOMES:
Correlation of blood pressure readings to rivaroxaban dosing | 48 hours
Correlation of blood pressure readings to symptomatology | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Roopen Arya, MBChB FRCP, Study Chair — King's College Hospital NHS Trust
Locations (1):
- Kings College Hospital NHS Foundation Trust, London, United Kingdom